CLINICAL TRIAL: NCT05247697
Title: Safety and Efficacy of Mirtazapine in the Treatment of Chronic Insomnia in Older Adults : The MIRAGE Study
Brief Title: Mirtazapine for Chronic Insomnia in Older Adults
Acronym: MIRAGE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Quebec Researchnetwork on aging (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20.105
Record Dates: First submitted 2022-01-12; First posted 2022-02-21 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Chronic Insomnia
Keywords: Insomnia; Mirtazapine; Aged
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mirtazapine

STUDY DESIGN:
Intervention Model Description: Prospective double blind placebo controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Mirtazapine 7.5 mg
  Interventions: Drug: Mirtazapine 7.5 MG Oral Tablet once daily at bedtime
- Control (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo oral tablet once daily at bedtime

INTERVENTIONS:
Drug: Mirtazapine 7.5 MG Oral Tablet once daily at bedtime — Mirtazapine 7,5 mg capsule
  Arms: Treatment
Drug: Placebo oral tablet once daily at bedtime — Matching placebo
  Arms: Control

SUMMARY:
Insomnia is highly prevalent in the older adult population. The pharmacolgical management of chronic insomnia includes benzodiazepines and Z-drugs (zolpidem, zopiclone). Although these drugs are indicated for insomnia, they are not without side effects. These drugs are associated with cognitive impairment, rebound insomnia, falls and addiction. Mirtazapine has a hypnotic and sedative effect related to the blocking of histamine-1 receptors. No clinical trials has evaluated the efficacy and safety of mirtazapine for insomnia in the older population.

The goal of the study is to assess the efficacy and safety of mirtazapine compared to a placebo in older adults with chronic insomnia.

This prospective double-blind placebo controlled trial will be conducted in adults 65 years and older with chronic insomnia. The treatment group will receive mirtazapine 7.5 mg at bedtime for 28 days and the control group will receive a matching placebo for 28 days. The sample size for the pilot study will be 60 subjects, 30 subjects in the treatment group and 30 subjects in the control group. The efficacy of mirtazapine will be measured using the Insomnia Severity Index and the Pittsburgh Sleep Quality Index. Safety will be monitored during the study

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* A report of sleep initiation or maintenance problems
* An adequate opportunity and circumstances to sleep,
* To have at least one daytime consequence in relation to sleep complaint.
* Sleep disorder and daytime consequences occur at least 3 times a week.
* Duration of sleep disorder and daytime consequences for at least 3 months
* Sleep complaint cannot be explained by a sleep disorder other than chronic insomnia.

Exclusion Criteria:

* Contrindication to mirtazapine
* Use of drug for insomnia
* Cognitive Behavioural Therapy for insomnia
* Use of Melatonin
* Active psychiatric illness
* Parkinson's disease
* Major Neurocognitive disorders
* More than one fall in the last 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | For Mirtazapine and placebo group : Assess the change in the Insomnia Severity Index between the initial examination (Day 1) and the end of the treatment course (Day 36)
  Self-reported insomnia symptoms using an insomnia severity scale from 0 to 28, 28 being the worst outcome
Pittsburgh Sleep Quality Index | For Mirtazapine and placebo group : Assess the change in the Pittsburgh Sleep Quality Index between the initial examination (Day 1) and the end of the treatment course (Day 36)
  Sleep scale from 0 to 21, 21 being the worst outcome

CONTACTS AND LOCATIONS:
Overall Officials: Patrick VQ Nguyen, Principal Investigator — Centre de Recerche du CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen PV, Dang-Vu TT, Forest G, Desjardins S, Forget MF, Vu TT, Nguyen QD, Kouassi E, Desmarais P. Mirtazapine for chronic insomnia in older adults: a randomised double-blind placebo-controlled trial-the MIRAGE study. Age Ageing. 2025 Mar 3;54(3):afaf050. doi: 10.1093/ageing/afaf050. PMID 40135470